CLINICAL TRIAL: NCT02054819
Title: A Pilot Study Treating Patients With Minimal Stage IV Non-Small Cell Lung Cancer (NSCLC) With Curative Intent
Brief Title: Treating NSCLC Minimal Stage IV With Curative Intent
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Didn't meet accrual goal, change in standard of care.
Sponsor: Leo W. Jenkins Cancer Center (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LJCC 2011-01
Record Dates: First submitted 2013-08-26; First posted 2014-02-04 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Other): Induction chemotherapy and concurrent radiation to primary tumor Cycle 1: irinotecan 65mg/m2 and cisplatin 30 mg/m2 on Day 1 and 8 Q 21 days Cycles 2-4: irinotecan 65 mg/m2, and cisplatin 30 mg/m2 Day 1 and 8 Q 21 days PLUS radiation therapy 66 Gy/7weeks/33 daily fractions
  Consolidation Radiation: therapy to metastatic sites At least 60 Gy total (taking into account a possible 3 Gy x 4 pre-treatment or equivalent) to all metastatic sites.
  Interventions: Other: Induction chemotherapy and concurrent radiation; Other: Consolidation: Radiation therapy to metastatic sites

INTERVENTIONS:
Other: Induction chemotherapy and concurrent radiation — Cycle 1: irinotecan 65mg/m2 and cisplatin 30 mg/m2 on Day 1 and 8 Q 21 days Cycles 2-4: irinotecan 65 mg/m2, and cisplatin 30 mg/m2 Day 1 and 8 Q 21 days PLUS radiation therapy 66 Gy/7weeks/33 daily fractions
Other: Consolidation: Radiation therapy to metastatic sites — At least 60 Gy total (taking into account a possible 3 Gy x 4 pre-treatment or equivalent) to all metastatic sites. For brain, 2.5 Gy x 14 to whole brain to follow stereotactic radiosurgery (SRS).

SUMMARY:
It is the hypothesis of this protocol that a subset of NSCLC patients with stage IVa disease can benefit from curative therapy and extends beyond the very limited subset of oligometastatic patients that have already been studied.

DETAILED DESCRIPTION:
In this study, patiently will be aggressively treated with 4 cycles of full dose platinum-based chemotherapy with concurrent radiation therapy to the primary tumor and identified mediastinal lymph nodal metastatic drainage. Local curative radiation will then target the oligometastatic tumor sites.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documented NSCLC, including squamous cell carcinoma, adenocarcinoma, large cell carcinoma including large cell neuroendocrine carcinoma and poorly differentiated (not otherwise specified - NOS) non-small cell lung cancer. Bronchial alveolar adenocarcinoma and totally resected tumors are excluded. All histology is to be reviewed at East Carolina University or designated participating center.
* Patients with Stage II-IIIB intra-thoracic disease with oligometastatic disease (hereafter referred to as "Stage IVa" disease) are eligible. Definition of Stage IVa:

Metastatic disease; either biopsy proven or with strong radiographic evidence suggesting its existence.

As determined by CT, MRI or PET no more than five distinct metastatic sites. All metastatic disease must be anatomically located in such a way as to permit a reasonable attempt at permanent ablation. Ablative measures may include surgery, stereotactic radiosurgery, and external beam therapy. Patients who meet the minimal metastatic disease requirement and who would otherwise have been staged II, IIIA or IIIB.

* Patients with tumors adjacent to a vertebral body are eligible as long as all gross disease can be encompassed in the radiation boost field.
* Patients must be ≥ 18 years of age.
* Patients with Zubrod (ECOG) performance status ≤ 2.
* Adequate hematologic function defined as: absolute neutrophil count (ANC) ≥ 1000/mm3, platelets ≥ 75,000/mm3, and hemoglobin ≥ 8 g/dL (prior to transfusions); adequate hepatic function defined as: total bilirubin ≤ 3.0 mg/dl, and adequate renal function defined as a serum creatinine level ≤ 2.0 mg/dl.
* Forced expiratory volume (FEV1) ≥ 800ml.
* Patients with weight loss < 20% over the past 3 months.
* Patients with a pleural effusion that is proven cytologically negative or is too small to tap.
* Women of childbearing potential must agree to practice effective contraception throughout the study plus four weeks.
* Pretreatment evaluations required for eligibility include:

A medical history, physical exam, and Zubrod performance status within 3 weeks prior to study entry.

Complete blodd count (CBC) with differential and platelet count, and laboratory profile must be completed within 3 weeks prior to study entry.

FEV1, CT scan of the chest or whole body PET (preferred), and a CT scan or MRI (preferred) of the brain within 4 weeks prior to study entry.

For women of childbearing potential, a serum or urine pregnancy test within a week prior to the start of protocol treatment.

Medical Oncology and Radiation Oncology consultation and approval.

* Patients must sign a study-specific consent form prior to study entry.

Exclusion Criteria:

* Prior systemic chemotherapy or radiotherapy that would interfere with delivery of treatment as outlined above as judged by the clinician.
* Cytologically malignant effusions.
* Metastatic disease beyond what is described in section 3.1.2.
* Active pulmonary infection not responsive to antimicrobial therapy.
* History of symptomatic interstitial pneumonitis.
* Significant symptomatic cardiac disease, i.e., unstable angina, uncompensated congestive heart failure, or uncontrolled cardiac ventricular arrhythmias.
* Patients with > grade 2 neuropathy.
* Evidence of malignancy in the past 2 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other in situ cancers.
* Women who are pregnant or breast feeding.
* Women of childbearing potential who are unwilling to practice effective contraception.
* Patients who currently are participating in other clinical trials and/or who have participated in other clinical trials in the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06; Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | Anticipated medial survival time is 8 - 10 months, however, all participants will be followed until death, assessed up to 100 months.
  Measure time of survival from enrollment to death from any cause, assessed up to 100 months.

SECONDARY OUTCOMES:
New metastatic disease | Anticipated time to progression is unknown, however, all patients will be followed for survival, up to 100 months.
  Measure of time from patient entry to time of new disease or progression of disease or date of death from any cause, whichever came first, assessed up to 100 months.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Walker, MD, PhD, Principal Investigator — Brody School of Medicine ar East Carolina University
Locations (1):
- Leo W. Jenkins Cancer Center, Greenville, North Carolina, United States